CLINICAL TRIAL: NCT03303963
Title: Culture Free Diagnosis and Follow-up of Multidrug Resistant Tuberculosis Patients
Brief Title: DIAgnostics for Multidrug Resistant Tuberculosis in Africa
Acronym: DIAMA
Status: Completed | Type: Observational
Sponsor: Dissou AFFOLABI (Other Government)
Collaborators: Rwanda Biomedical Centre (Other); The Tuberculosis Reference Laboratory Bamenda (Unknown); Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Jimma University (Other); Service de Pneumophtisiologie, Hôpital Ignace Deen (Unknown); University of the Sciences, Techniques and Technologies of Bamako (Other); Damien Foundation (Other); Cheikh Anta Diop University, Senegal (Other); Institute of Tropical Medicine, Belgium (Other); World Health Organization (Other); London School of Hygiene and Tropical Medicine (Other); Genoscreen (Other)
Responsible Party: Sponsor-Investigator, Dissou AFFOLABI, Professor (Deputy Head of the Laboratory), Laboratoire de Référence des Mycobactéries
Organization: Laboratoire de Référence des Mycobactéries (Other Government)
Other Study IDs: DRIA2014-326
Record Dates: First submitted 2017-09-24; First posted 2017-10-06 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Tuberculosis, Multidrug-Resistant
Keywords: culture-free; tuberculosis; multidrug resistant; diagnosis; follow-up; africa; molecular tools
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis; Disease | interventions — Microscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum.
  At the enrolment, three samples (spot-overnight-spot) will be collected for the comparison of phenotypic results against molecular results.
  During the treatment, two monthly samples (overnight-spot) will be collected for the comparison of culture result against FDA Microscopy and GeneXpert Ct values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rifampicin resistant and susceptible patients: Study 1: Patients detected positive by the GeneXpert Mycobacterium tuberculosis/Rifampicin (susceptible and resistant to rifampicin)
  Interventions: Diagnostic Test: Deeplex test, MolBio TrueNat for 2nd line, GeneXpert 2nd line
- Rifampicin resistant patients: Study 2: Follow up of the rifampicin resistant patients included in the study 1 during their treatment
  Interventions: Diagnostic Test: Fluorescein DiAcetate (FDA) Microscopy,GeneXpert Ct value, pre-rRNA synthesis

INTERVENTIONS:
Diagnostic Test: Deeplex test, MolBio TrueNat for 2nd line, GeneXpert 2nd line — Improvement of the diagnosis of Multi Drug Resistant-Tuberculosis patients with culture-free approaches. We have planned to diagnose Tuberculosis resistance to 1st and 2nd line drugs through novel molecular multiplex assays (Study 1) by:
  * Validating the Deeplex test and establish a network for shipment of sputum samples in ethanol to regional reference laboratories (Study 1 - phase 1)
  * Validating the Molbio Truenat test as a point of care test (Study 1 - phase 2)
  * Validating the Cepheid GeneXpert 2nd line cartridge at the district level (Study 1 -phase2)
  Groups: Rifampicin resistant and susceptible patients
Diagnostic Test: Fluorescein DiAcetate (FDA) Microscopy,GeneXpert Ct value, pre-rRNA synthesis — Improvement of the management of Multi Drug Resistant-Tuberculosis patients with culture-free approaches. We have planned to set up alternative culture-free approaches for the monitoring of patients' response to Multi Drug Resistant-Tuberculosis treatment (Study 2), with:
  * FDA microscopy
  * Measurement of bacterial load by following Cycle threshold (Ct) values in GeneXpert Mycobacterium tuberculosis/Rifampicin
  * Measurement of pre-rRNA synthesis
  Groups: Rifampicin resistant patients

SUMMARY:
Recent advances in molecular diagnostics of tuberculosis, especially the GeneXpert Mycobacterium tuberculosis/Rifampicin test have reduced the time to diagnose Rifampicin Resistant Tuberculosis (RR-TB) but only rifampicin resistance is diagnosed, leading to presumptive diagnosis of resistance to isoniazid and maybe other drugs. Thus in low and middle income countries, most drug sensitivity testing relies on phenotypic drug resistance testing, which takes up to 4 months. In addition, currently, culture on monthly sputum samples is recommended by the World Health Organization for follow-up of Rifampicin Resistant Tuberculosis patients under treatment. Unfortunately, culture is often not locally available and samples need to be transported from field to culture laboratories. The associated transport delays lead to high rates of contamination and false negative culture, particularly in laboratories in low resource settings. Many gaps for the diagnosis and management of RR-TB patients still need to be addressed and the DIAMA project (DIAgnostics for Multidrug resistant tuberculosis in Africa) study aims to address some of them.

DETAILED DESCRIPTION:
The proposed DIAMA (DIAgnostics for Multidrug resistant tuberculosis in Africa) study aims to address current gaps in the diagnosis and management of patients with Multi-Drug-Resistant (MDR) tuberculosis. Building on existing networks and research collaborations previously funded by the European & Developing Countries Clinical Trials Partnership (EDCTP), this project involved partners in West, Central, and East Africa. It aims to evaluate and implement rapid and accurate molecular tests for several anti Tuberculosis drugs, to replace the current dependency on phenotypic drug resistance testing, which takes up to 4 months and is technically so demanding that few laboratories can perform it correctly.

The project builds on the continuous surveillance of Tuberculosis retreatment patients for rifampicin resistance. Two African partners (Benin and Rwanda) with advanced molecular laboratories are establishing reference laboratories for the 'Deeplex' assay, a novel multiplex deep sequencing-based drug resistance diagnostic platform that simultaneously provides sequence information of genes that confer resistance to several key anti tuberculosis drugs. Partners are recruiting all patients with rifampicin resistant Tuberculosis, and a subset of those with rifampicin sensitive Tuberculosis. In a first phase, sputum will be shipped for the Deeplex assay, for comparison against phenotypic DST, the reference method for detecting resistance to 1st and 2nd line drugs. In addition, since Whole Genome Sequencing is the "reference" of molecular tests, Deeplex assay will also be validated again this test. In a second phase, Cepheid 2nd line Xpert and Molbio Truenat test, two 'lower tech' tests at the last stages of laboratory validations, will also be validated. The Cepheid Xpert 2nd line cartridge can be implemented in existing Xpert machines used for the Xpert MTB/Rif assays. These tests will be compared versus the Deeplex assay and versus WGS

Using the latest advances in DataTocare software developed by one of the project partners, molecular results will be communicated in real time to the National Tuberculosis Programmes, so that Multi Drug Resistant Tuberculosis patients can swiftly start appropriate treatment. The added-value of this system will be evaluated as a pilot study in some sites.

Lastly, once patients have initiated MDR treatment, they will be monitored for treatment success by faster alternative approaches to the WHO recommended monthly cultures: serial sputum samples will have Fluorescein DiAcetate (FDA) vital stain microscopy, measurement of the bacterial load using the Xpert MTB/Rif as well as precursor of ribosomal RNA measurement (pre-rRNA).

Together, these advances are expected to dramatically improve the currently dismal prognosis of MDR-TB in health systems in resource-poor settings.

ELIGIBILITY:
Inclusion criteria:

* Being ≥ 15 year old
* Having a positive test on GeneXpert (M. tuberculosis) with or without resistance detected to rifampicin
* Willing and able to provide written informed consent, or for minors: assent from and consent from a legal representative

Exclusion Criteria: None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Two multi center observational studies will be conducted:
  Study 1: Cross sectional study for Tuberculosis(TB) cases aged ≥ 15 (all Rifampicin resistant (RR) ones (new cases or retreatment patients) and equal number of Rifampicin sensitive retreatment patients from the same country) with comparison of TB resistance diagnostic test performance at baseline. There are 2 phases in this project; phase 1 is the comparison of Deeplex results against the phenotypic results and WGS (Gold standard), phase 2 is the comparison of MolBio TrueNat and GeneXpert 2nd generation results against Deeplex and WGS (gold standard).
  Study 2: Cohort study of RR-TB patients (recruited in Study 1) under treatment with comparison of the performance of FDA and GeneXpert compared to solid culture
Sampling Method: Non-Probability Sample
Enrollment: 3356 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Validation of Deeplex test | 4 years
  Concordance between phenotypic Drug Susceptibility Test, WGS and Deeplex results
Validation of GeneXpert 2nd line | 4 years
  Concordance between WGS, Deeplex results and GeneXpert 2nd line results
Validation of MolBio TrueNat for INH, FQ and BDQ | 4 years
  Concordance between WGS, Deeplex results and MolBioTrueNat results
Validation of FDA microscopy | 4 years
  Concordance between Culture results and FDA microscopy results
Validation of GeneXpert Ct value | 4 years
  Concordance between Culture results and GeneXpert Ct value results

SECONDARY OUTCOMES:
Estimation of proportion of additional resistance in patients resistant to Rifampicin | 4 years
  Evaluation to be done with the Deeplex test
Measurement of the association of specific mutations against some drugs with programmatic treatment outcome | 4 years
  Evaluation to be done with the Deeplex test
Evaluation of the add value of Connectivity system in the management of Multi Drug Resistant-Tuberculosis patients | 2 years
  Evaluation to be done with Data2Care connectivity system

CONTACTS AND LOCATIONS:
Overall Officials: Dissou AFFOLABI, MD, MSc, PhD, Principal Investigator — Laboratoire de Référence des Mycobactéries
Locations (10):
- Institute of Tropical Medecine, Antwerp, Belgium
- Centre National Hospitalier Universitaire de Pneumo-Phtisiologie de Cotonou, Cotonou, Atlantique/Littoral, Benin
- The Tuberculosis Reference Laboratory Bamenda, Bamenda, Cameroon
- Institut National de Recherche Biomédicale (INRB), Kinshasa, Democratic Republic of the Congo
- Jimma University, Jīma, Ethiopia
- Service de Pneumophtisiologie, Hôpital Ignace Deen, Conakry, Conakry, Guinea
- Université des Sciences, des Techniques et des Technologies de Bamako, SEREFO, Bamako, Mali
- Damien Fundation, Ibadan, Nigeria
- Rwanda Biomedical Center (RBC), Kigali, Rwanda
- Université Cheick Anta Diop (UCAD), Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boehme CC, Nabeta P, Hillemann D, Nicol MP, Shenai S, Krapp F, Allen J, Tahirli R, Blakemore R, Rustomjee R, Milovic A, Jones M, O'Brien SM, Persing DH, Ruesch-Gerdes S, Gotuzzo E, Rodrigues C, Alland D, Perkins MD. Rapid molecular detection of tuberculosis and rifampin resistance. N Engl J Med. 2010 Sep 9;363(11):1005-15. doi: 10.1056/NEJMoa0907847. Epub 2010 Sep 1. PMID 20825313
- [Result] Bastos ML, Hussain H, Weyer K, Garcia-Garcia L, Leimane V, Leung CC, Narita M, Pena JM, Ponce-de-Leon A, Seung KJ, Shean K, Sifuentes-Osornio J, Van der Walt M, Van der Werf TS, Yew WW, Menzies D; Collaborative Group for Meta-analysis of Individual Patient Data in MDR-TB. Treatment outcomes of patients with multidrug-resistant and extensively drug-resistant tuberculosis according to drug susceptibility testing to first- and second-line drugs: an individual patient data meta-analysis. Clin Infect Dis. 2014 Nov 15;59(10):1364-74. doi: 10.1093/cid/ciu619. Epub 2014 Aug 5. PMID 25097082
- [Result] Aung KJ, Van Deun A, Declercq E, Sarker MR, Das PK, Hossain MA, Rieder HL. Successful '9-month Bangladesh regimen' for multidrug-resistant tuberculosis among over 500 consecutive patients. Int J Tuberc Lung Dis. 2014 Oct;18(10):1180-7. doi: 10.5588/ijtld.14.0100. PMID 25216831
- [Result] Piubello A, Harouna SH, Souleymane MB, Boukary I, Morou S, Daouda M, Hanki Y, Van Deun A. High cure rate with standardised short-course multidrug-resistant tuberculosis treatment in Niger: no relapses. Int J Tuberc Lung Dis. 2014 Oct;18(10):1188-94. doi: 10.5588/ijtld.13.0075. PMID 25216832
- [Result] Van Deun A, Maug AK, Salim MA, Das PK, Sarker MR, Daru P, Rieder HL. Short, highly effective, and inexpensive standardized treatment of multidrug-resistant tuberculosis. Am J Respir Crit Care Med. 2010 Sep 1;182(5):684-92. doi: 10.1164/rccm.201001-0077OC. Epub 2010 May 4. PMID 20442432
- [Derived] Inbaraj LR, Daniel J, Sathya Narayanan MK, Srinivasalu VA, Bhaskar A, Scandrett K, Rajendran P, Kirubakaran R, Shewade HD, Malaisamy M, Padmapriyadarsini C, Takwoingi Y. Truenat MTB assays for pulmonary tuberculosis and rifampicin resistance in adults and adolescents. Cochrane Database Syst Rev. 2025 Mar 24;3(3):CD015543. doi: 10.1002/14651858.CD015543.pub2. PMID 40122135
- [Derived] Pillay S, Steingart KR, Davies GR, Chaplin M, De Vos M, Schumacher SG, Warren R, Theron G. Xpert MTB/XDR for detection of pulmonary tuberculosis and resistance to isoniazid, fluoroquinolones, ethionamide, and amikacin. Cochrane Database Syst Rev. 2022 May 18;5(5):CD014841. doi: 10.1002/14651858.CD014841.pub2. PMID 35583175

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT03303963/Prot_SAP_ICF_000.pdf